CLINICAL TRIAL: NCT04352036
Title: Constitution of a Prospective Cohort of Patients With Acute Suppurative Hidrosadenitis Followed in the Great West: the COVER Cohort (Verneuil Cohort)
Acronym: COVER
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0418
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Acute Hidrosadenitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skin biopsies and bacteriological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patient
  Interventions: Other: no interventional study

INTERVENTIONS:
Other: no interventional study — no interventional study

SUMMARY:
Our primary objective with this cohort will be to define the different phenotypes of acute hidrosadenitis, the characterization of which is essential to define suitable therapeutic approaches. Indeed, our recent data allow us to note that there would be different phenotypes of acute hidrosadenitis and therefore different pathologies inducing different follow-ups and care.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with acute hidrosadenitis by a dermatologist
* Patient agreeing to be part of the study

Exclusion Criteria:

* Major under guardianship
* Protected persons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population studied will relate to patients consulting or being hospitalized for Acute Hidrosadenitis, whatever its severity.
Sampling Method: Probability Sample
Enrollment: 465 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2030-02-20 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
Description of the natural history and identification of the different clinical forms of acute hidrosadenitis | through study completion, an average of 3 years
  history of the disease, classification of Hurley, Canoui-Poitrine and van der Zee and Jemec
Prevalence of severe forms (grade II, III) | through study completion, an average of 3 years
  Number of patients with severe disease (grades II and III)
Definition of different phenotypes of acute hidrosadenitis | through study completion, an average of 3 years
  patient history, Canoui-Poitrine and van der Zee and Jemec classification, blood and urine tests, imaging
Identify the environmental factors associated with the chronicity of the disease | through study completion, an average of 3 years
  socio-demographic data
Identify the environmental factors associated with the chronicity of the disease | through study completion, an average of 3 years
  questionnaire for collecting dietary habits
Identify the environmental factors associated with the chronicity of the disease | through study completion, an average of 3 years
  biological nutritional assessment research for a dysmetabolic syndrome
Identify the environmental factors associated with the chronicity of the disease | through study completion, an average of 3 years
  research for a dysmetabolic syndrome
Identify the environmental factors associated with the chronicity of the disease | through study completion, an average of 3 years
  lifestyle questionnaire assessing the impact on quality of life

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - Chru Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH, Le Mans
  - CH bretagne sud, Lorient
  - CHU de Nantes - Dermatologie, Nantes
  - Chr D'Orléans, Orléans
  - CHU Milétrie, Poitiers
  - Ch de Cornouaille, Quimper
  - CHU Pontchaillou, Rennes
  - Ch Saint-Brieuc, Saint-Brieuc
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided